CLINICAL TRIAL: NCT04673656
Title: Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study to Evaluate the Effect of BKR-017 on Insulin Resistance and Other Metabolic Parameters in Type 2 Diabetes Patients
Brief Title: Dose-Response Study to Evaluate the Effect of BKR-017 on Insulin Resistance and Other Metabolic Parameters in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioKier Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CL-501
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group 1 (Placebo Comparator): Group 1 will receive 84 days of placebo BID
  Interventions: Dietary Supplement: BKR-017
- Test Group 2 (Active Comparator): Group 2 will receive 84 days of 0.5 g of BKR-017 BID
  Interventions: Dietary Supplement: BKR-017
- Test Group 3 (Active Comparator): Group 3 will receive 84 days of 1.0 g of BKR-017 BID
  Interventions: Dietary Supplement: BKR-017
- Test Group 4 (Active Comparator): Group 4 will receive 84 days of 1.5 g of BKR-017 BID
  Interventions: Dietary Supplement: BKR-017

INTERVENTIONS:
Dietary Supplement: BKR-017 — Nutrient butyrate into a colon-targeted tablet formulation (BKR-017) is intended to stimulate secretion of GLP-1 from L-cells in the lower gut. Butyrate delivered to the colon in tablet form will not cause the side-effects seen with formation of butyrate by fermentation.
  Other Names: Butyrate

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, dose-response study of BKR-017 and placebo that will be conducted at two investigative sites. The total duration of subject involvement is approximately 15 weeks; the screening period can be up to 3 weeks prior to the start of test period, followed by a 12-week test period. During the test period, subjects will self-administer three tablets of test product, two times daily: before breakfast and before bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 70 years at the time of screening, inclusive
* Diagnosed with T2D and under the care of a healthcare professional for its management, or newly diagnosed (as participant in the study) with T2D
* HbA1c 6.5% -10.5%, inclusive
* Has given written informed consent to participate in this study
* Willing to complete 84-day test period
* Willing to maintain current diet and exercise routine and current prescription medications for the duration of the study

Exclusion Criteria:

* Type 1 diabetes
* History of bariatric or intestinal surgery
* Active gastrointestinal disease including but not limited to irritable bowel syndrome, inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis), diverticulitis, gastroparesis
* Active and clinically significant hepatic, pancreatic disease, or renal disease as determined by the investigator
* History of heart disease that in the opinion of the investigator should exclude the subject from the study
* Severely uncontrolled hypertension at screening defined as a systolic blood pressure > 180 mmHg or a diastolic blood pressure > 110 mmHg on the average of two seated measurements after being at rest for at least 5 minutes
* Untreated or uncontrolled hyperthyroidism or hypothyroidism, or other significant thyroid disease
* Active significant infection as determined by the investigator
* Known allergy to butyrate or any of the components of the tablets
* Subjects planning to make major changes to diet and physical activity during the trial duration
* Participation in a clinical trial and/or treatment with an investigational drug during the 30 days before screening, or within 5 half-lives of receipt of an investigational drug or twice the duration of the biological effect of any investigational drug (whichever is longer)
* Pregnant, nursing, or trying to become pregnant
* In the investigator's judgment, the subject is not suitable for the study for any other reason or cannot commit to the requirements of the study.
* Subject is taking one or more of the excluded therapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Changes in HOMA-IR | Baseline, Day 1, during the treatment period at days 21, 42, and 63, and at end of treatment period, Day 84
  Changes in HOMA-IR at Days 21, 42, 63, and 84 using repeated measures ANCOVA

SECONDARY OUTCOMES:
Changes in fasting low-density lipoprotein-cholesterol (LDL-C) | Baseline, Day 1, during the treatment period at day 42, and at end of treatment period, Day 84
  Changes in fasting low-density lipoprotein-cholesterol (LDL-C) at Days 1, 42, and 84
Changes in fasting triglycerides | Baseline, Day 1, during the treatment period at days 42, and at end of treatment period, Day 84
  Changes in fasting triglycerides at Days 1, 42, and 84
Changes in HbA1c | Baseline, Day 1, during the treatment period at day 42, and at end of treatment period, Day 84
  Changes in HbA1c at Days 1, 42, and 84
Changes in fasting glucose | Baseline, Day 1, during the treatment period at day 42, and at end of treatment period, Day 84
  Changes in fasting glucose at Days 1, 42, and 84
Changes in fasting insulin | Baseline, Day 1, during the treatment period at day 42, and at end of treatment period, Day 84
  Changes in fasting insulin at Days 1, 42, and 84

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Duke Clinical Research at Pickett Road, Durham, North Carolina
  - Duke Clinical & Translational Science Institute (CTSI), Kannapolis, North Carolina